CLINICAL TRIAL: NCT02340910
Title: Dose-Response Effects of Whole Body Vibration on Spasticity and Walking in SCI
Acronym: WBV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shepherd Center, Atlanta GA (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WBV-612299
Record Dates: First submitted 2015-01-09; First posted 2015-01-19 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Spinal Cord Injury
Keywords: spasticity; whole body vibration; walking
MeSH Terms: conditions — Spinal Cord Injuries; Muscle Spasticity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Masked allocation and intervention
Oversight: Data Monitoring Committee: No

ARMS (2):
- Short duration (Experimental): Short Duration WBV consists of 8 45-sec bouts of 50Hz WBV followed by a 1-minute seated rest
  Interventions: Procedure: Short Duration
- Long duration (Experimental): Long Duration WBV consists of 16 bouts 45-sec of 50Hz WBV followed by a 1-minute seated rest
  Interventions: Procedure: Long Duration

INTERVENTIONS:
Procedure: Short Duration — During each WBV repetition, subjects will stand on the vibration platform of the WBV device with knees slightly bent (approximately 30 degrees flexion). The subject will hold the handrails for balance and the WBV device will be turned on. The subject will receive a total of 6 minutes of WBV at a frequency of 50 Hz.
  Arms: Short duration
Procedure: Long Duration — During each WBV repetition, subjects will stand on the vibration platform of the WBV device with knees slightly bent (approximately 30 degrees flexion). The subject will hold the handrails for balance and the WBV device will be turned on. The subject will receive a total of 12 minutes of WBV at a frequency of 50 Hz.
  Interventions will occur for a total of 20 sessions over 4 consecutive weeks .
  Arms: Long duration

SUMMARY:
This study will enroll people with SCI who have spasticity and some ability to walk. The goal is to understand if standing on a platform and receiving WBV results in decreased spasticity and improved walking ability. Published article is available (PMID: 29959653)

DETAILED DESCRIPTION:
Phase 1 of this study has been successfully completed. The results of Phase 1 indicate that a single session of WBV lasting for a total of 6 minutes (delivered in eight 45-sec bouts) at a high-frequency (50Hz) was associated with the largest decrease in spasticity (as measured by the pendulum test). The goal for Phase 2 is to determine whether longer doses of WBV result in greater reductions in spasticity as well as improvements in walking ability. Two different doses of WBV, a short dose and a long dose, will be tested.

ELIGIBILITY:
Inclusion Criteria: have spinal cord injury of at least 6 months duration; be between the ages of 16 - 72 years old; be able to sit at the edge of the mat without the assistance of another person; be able to tolerate standing; have at least mild spasticity affecting the lower extremity muscles; be able to understand and provide own consent; you may participate if you use prescription medications, including baclofen pump for control of spasticity, as the dosage is stable; obtain medical clearance for standing if you have been injured more than 1 year and are not regularly walking or standing.

Exclusion Criteria: progressive or potentially progressive spinal lesions, including degenerative, or progressive vascular disorders of the spine and/or spinal cord; neurologic level below spinal level T12; history of cardiovascular irregularities; problems following instructions; orthopedic problems that would limit your participation in the protocol (e.g. knee or hip flexion contractures of greater than 10 degrees)

Ages: 16 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2015-02-02 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Spasticity Assessments | Estimated 1 hour
  Pendulum test, Spinal Cord Injury Spasticity Evaluation Tool (SCI-SET) Questionnaire, Electrophysiological testing (Soleus H-reflex)

SECONDARY OUTCOMES:
Walking ability | Estimated 30 minutes
  Walking speed, endurance and pattern will be assessed while wearing motion capture sensors
Strength | Estimated 20 minutes
  5 times sit to stand assessment, testing of upper leg muscle strength using force measurements
Pain perception | Estimated 20 minutes
  SCI Pain Basic Dataset Questionnaire
Upper Extremity Tests | Estimated 5 minutes
  For participants who have a cervical level of injury, pinch strength will be measured using a hand-held device and the nine-hole peg test will be used to measure hand function.
Ankle Clonus Test/Foot | Estimated 15 minutes
  Ankle spasticity will be measured using motion capture sensors to record ankle joint angles.

CONTACTS AND LOCATIONS:
Locations (1):
- Shepherd Center, Inc., Atlanta, Georgia, United States

REFERENCES:
- [Background] Estes S, Iddings JA, Ray S, Kirk-Sanchez NJ, Field-Fote EC. Comparison of Single-Session Dose Response Effects of Whole Body Vibration on Spasticity and Walking Speed in Persons with Spinal Cord Injury. Neurotherapeutics. 2018 Jul;15(3):684-696. doi: 10.1007/s13311-018-0644-1. PMID 29959653
- See also: Related Info — http://shepherd.org